CLINICAL TRIAL: NCT03025100
Title: Adherence to Venous Thromboembolism Prophylaxis Guidelines in Hospitalized Elders
Brief Title: VTE Prophylaxis Guidelines in Hospitalized Elders
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Hartford Foundation (Other); National Institute on Aging (NIA) (NIH); T. Franklin Williams Scholars (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00056253; R03AG048007-01 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prospective: A sample of 120 patients aged 60 years or older admitted to General Medicine at Duke University Hospital will be enrolled in the prospective cohort study. A convenience sample will be derived from a randomized daily list of general medicine admissions; weekend admissions will be excluded as these patients will not be captured within 24 hours of hospital admission.

SUMMARY:
Guideline directed use of pharmacologic Venous thromboembolism (VTE) prophylaxis emphasizes mobility evaluation. Mobility is a key component of risk stratification. Poor mobility evaluation by providers may be a significant barrier to appropriate use of VTE prophylaxis. The investigators aim is to propose to determine whether level of mobility during hospitalization is being used to influence use and duration of VTE prophylaxis among medically ill hospitalized elders. To achieve this aim, the investigator will collect prospective observational data to objectively measure inpatient mobility using patient mounted accelerometers during patient hospital stays.

The investigator's goal is to improve the appropriateness of use of VTE prophylaxis among those in which the risks of harm may outweigh the benefit. Results from this study will provide important insights about use of risk assessment, and the relationship between patient mobility and VTE prophylaxis. These results are critical to understanding how to take the next steps toward improving the appropriate use and safety of anticoagulants in hospitalized older adults. Information from this study could be used in future proposals to study interventions to ultimately improve hospital practice in the care of older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 60 or older
2. Admitted to General Medicine at Duke University

Exclusion Criteria:

1. Clear contraindications to pharmacologic VTE prophylaxis
2. Receiving surgery during their index hospital stay
3. On observation admission status
4. On negative pressure room respiratory isolation
5. Wrist site is not available, i.e. wearing bilateral wrist IVs, skin breakdown at the time of screening
6. Ankle site is not available, i.e. patients with leg ulcer at the time of screening
7. Lacking decision-making ability (such as from severe cognitive impairment) and no LAR available
8. Non-English speakers

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of patients aged 60 years or older admitted to General Medicine at Duke University Hospital will be enrolled in a prospective cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03-04 (Actual); Study Completion 2017-03-04 (Actual)

PRIMARY OUTCOMES:
Total number of minutes of activity (using objective accelerometer data). | Length of hospital stay or up to 7 days during the patient's hospital stay.
Total number of minutes of inactivity (using objective accelerometer data). | Length of hospital stay or up to 7 days during the patient's hospital stay.

SECONDARY OUTCOMES:
Total number of steps (using objective accelerometer data). | Length of hospital stay or up to 7 days during the patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Juliessa Pavon, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States